CLINICAL TRIAL: NCT00554671
Title: Group Intervention for DM Guideline Implementation
Brief Title: Pharmacist-led Group Medical Visits to Help With Diabetes Management
Acronym: MEDIC-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IAB 06-269
Record Dates: First submitted 2007-11-05; First posted 2007-11-07 (Estimated); Results first posted 2014-12-31 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Diabetes Mellitus; Cardiovascular Diseases
Keywords: Diabetes Mellitus; Clinical pharmacists; guideline adherence; group medical visits; behavioral modification; pharmacotherapy
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases | interventions — Self-Help Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pharmacist-led Group Visits (Experimental): Algorithm driven medication titration, Behavioral: Monitoring, Behavioral: Group support, Behavioral: Self efficacy
  Interventions: Other: Algorithm driven medication titration; Behavioral: Monitoring; Behavioral: Group support; Behavioral: Self efficacy
- Usual Care (No Intervention): Patient continues on usual care for diabetes

INTERVENTIONS:
Other: Algorithm driven medication titration — Clinical pharmacists will change medications to achieve goals in hypertension, dyslipidemia and diabetes
  Arms: Pharmacist-led Group Visits
Behavioral: Monitoring — Clinical pharmacists will monitor the progress of patients in lifestyle modification and cardiac risk factor control goals
  Arms: Pharmacist-led Group Visits
Behavioral: Group support — Peer support are provided in the group setting
  Arms: Pharmacist-led Group Visits
Behavioral: Self efficacy — Patients are taught with self-monitoring skills for diabetes and blood pressure, as well as healthy cooking and practiced under supervision
  Arms: Pharmacist-led Group Visits

SUMMARY:
This is a multi-site open label randomized controlled study of patients with type 2 diabetes undergoing pharmacist-led group medical visits that include education by a multi-disciplinary personnel, behavioral modification and pharmacotherapy case management vs. usual care

DETAILED DESCRIPTION:
Project Background: Diabetes, hypertension, and dyslipidemia are chronic diseases that can lead to heart attack and stroke, and require interventions at patient and organizational levels to promote sustainable lifestyle and medication changes for cardiac risk reduction that are costly. Group intervention has emerged as a potentially cost-saving patient-centered approach to help achieve the necessary lifestyle and medication changes for the treatment of some chronic diseases, but its efficacy in absence of direct physician participation is not well demonstrated in diabetes. Our preliminary data have shown that our pharmacist-based, group diabetes management program at the Providence VAMC has achieved significant improvements in glycemic control and variable success toward improvement in blood pressure and lipid control in type 2 diabetic patients, through education, behavioral intervention and aggressive pharmacotherapy in 4 weekly group sessions. However, we do not know the long-term sustainability of this intervention, the exportability, the costs to the VA and the health-related quality-of-life implications of patients enrolled in our programs.

Project Objectives: To assess whether a non-physician-based, group diabetes behavioral and pharmacotherapy intervention program for 12 months will: 1. improve cardiac risk factors, 2. improve health-related quality-of-life, 3. add only minimal institutional cost; when compared to usual care in veterans with type 2 diabetes.

Project Methods: We propose a 3-site randomized-controlled study to test the efficacy of a pharmacist-based, group diabetes behavioral and pharmacotherapy intervention program (treatment arm) for 13 months vs. usual care (control arm) in achieving cardiac risk reduction in type 2 diabetic patients with Hemoglobin A1c >7% and at least one other cardiac risk factor such as smoking, hyperlipidemia or hypertension not at national guideline recommended goals. The interventions in the treatment arm will consist of two phases. Phase 1 (intensive intervention) consists of weekly group sessions of education by a nurse, a physical therapist, and a dietician; and behavioral modification and medication titration by a clinical pharmacist targeting the control of glycemia, smoking, blood pressure, and lipids for 4 weeks. Phase 2 consists of quarterly booster sessions for 1 year to prevent relapse. Patients in the control arm will continue on usual care. Our study endpoints will be the difference between the 2 groups after 13 months of study enrollment in: 1) hemoglobin a1c, blood pressure, LDL cholesterol and smoking 2) health-related quality of life (SF-36V) scores, and 3) healthcare costs from the VA perspective. A total of 250 patients will be enrolled from 3 VAMC sites and followed for 13 months.

ELIGIBILITY:
Inclusion Criteria:

Diabetic veterans with HbA1c >7.0% and at least one of the following:

* being a smoker (any cigarette smoking < 30 days)
* having an LDL >100 mg/dl or a blood pressure >130/80 mm Hg documented in at least two occasions within the last 6 months
* able to participate and discuss their DM and cardiac risk control in a group setting and sign informed consent

Exclusion Criteria:

* patients without eligible cardiac risk factors within the last 6 months
* those who are unable to attend the group sessions
* or disease conditions such as psychiatric instability (acutely suicidal, psychotic) or organic brain injury that preclude them from performing DM self-care
* patients with conditions that would preclude them from standard algorithm-based medication dose titrations such as those who are pregnant or with complex co-morbidities as defined by New York Heart Association Class 3 or 4 heart failure, liver cirrhosis, end-stage renal disease on dialysis and end-stage cancer will be excluded from the study
* all women of childbearing age will have a pregnancy test before study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2008-05; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Chih H Wu, MD, Principal Investigator — Providence VA Medical Center, Providence, RI
Locations (3):
- United States (3):
  - VA Connecticut Health Care System (West Haven), West Haven, Connecticut
  - VA Pacific Islands Health Care System, Honolulu, Honolulu, Hawaii
  - Providence VA Medical Center, Providence, RI, Providence, Rhode Island

REFERENCES:
- [Background] Taveira TH, Pirraglia PA, Cohen LB, Wu WC. Efficacy of a pharmacist-led cardiovascular risk reduction clinic for diabetic patients with and without mental health conditions. Prev Cardiol. 2008 Fall;11(4):195-200. doi: 10.1111/j.1751-7141.2008.00008.x. PMID 19476571
- [Derived] Wu WC, Taveira TH, Jeffery S, Jiang L, Tokuda L, Musial J, Cohen LB, Uhrle F. Costs and effectiveness of pharmacist-led group medical visits for type-2 diabetes: A multi-center randomized controlled trial. PLoS One. 2018 Apr 19;13(4):e0195898. doi: 10.1371/journal.pone.0195898. eCollection 2018. PMID 29672567

RESULTS

PARTICIPANT FLOW:
Groups:
- Pharmacist-led Group Medical Visits: Pharmacist-led group medical visits which consists of medication titration and behavioral modification
  Algorithm driven medication titration: Clinical pharmacists will change medications to achieve goals in hypertension, dyslipidemia and diabetes
  Monitoring: Clinical pharmacists will monitor the progress of patients in lifestyle modification and cardiac risk factor control goals
  Group support: Peer support are provided in the group setting
  Self efficacy: Patients are taught with self-monitoring skills for diabetes and blood pressure, as well as healthy cooking and practiced under supervision
- Usual Care: Patients continued on usual care without pharmacist-led group medical visits
Period: Overall Study
Arm/Group | Pharmacist-led Group Medical Visits | Usual Care
Started | 117 | 133
Completed | 97 | 117
Not Completed | 20 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pharmacist-led Group Medical Visits | Usual Care | Total
Number analyzed (Participants) | 117 | 133 | 250
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (8.7) | 65.0 (9.8) | 65.4 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 128 | 240
  Male | 5 | 5 | 10
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 88 | 104 | 192
  African American | 12 | 15 | 27
  Asian Pacific Islander | 15 | 8 | 23
  Hispanic | 0 | 4 | 4
  Unknown | 2 | 2 | 4
Hemoglobin A1c [Mean (Standard Deviation); unit: percent Hemoglobin A1c] | 8.2 (1.5) | 8.2 (1.3) | 8.2 (1.4)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 136.5 (19.0) | 136.2 (17.4) | 136.3 (18.1)
LDL cholesterol [Mean (Standard Deviation); unit: mg/dL] | 87.6 (29.8) | 93.7 (33.7) | 91.0 (32.1)

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1c
Description: Hemoglobin A1c levels at 6 months
Time Frame: 6 months
Population: At the 6 month visit, some patients dropped out of the study or died.
Measure: Mean (Standard Deviation); unit: percent Hemoglobin A1c
Arm/Group | Pharmacist-led Group Medical Visits | Usual Care
Number analyzed (Participants) | 102 | 122
percent Hemoglobin A1c | 7.8 (1.2) | 8.1 (1.4)

2. Primary Outcome: Hemoglobin A1c
Description: hemoglobin A1c levels at 13 months
Time Frame: 13 months
Measure: Mean (Standard Deviation); unit: percent Hemoglobin A1c
Arm/Group | Pharmacist-led Group Medical Visits | Usual Care
Number analyzed (Participants) | 97 | 117
percent Hemoglobin A1c | 7.9 (1.3) | 8.0 (1.4)

3. Secondary Outcome: Change From the Baseline in the Hr-QOL as Assessed by SF-36V at 13 Months of Study Enrollment
Description: Medical Outcomes Study 36-Item Short Form Survey (SF-36) is a popular, multi-purpose health status survey that addresses quality of life from physical and mental health perspectives. SF-36v is the survey adapted for veterans. Items are summed and averaged in two subscores, the Physical Composite Summary Score and the Mental Composite Summary Score, and scaled to a range of 0 to 100, with lower scores denoting poorer health.
Time Frame: Baseline and 13 months
Population: 117 patients randomized to Pharmacist-led Group Medical Visits, 2 patients died before study end date and 18 patients dropped out.133 patients randomized to Usual care, 4 patients died before study end date and 12 patients dropped out.
Measure: Mean (Standard Deviation); unit: Scores of SF-36v
Groups:
- Pharmacist-led Group Visits: Pharmacist-led group medical visits which consists of medication titration and behavioral modification
  Algorithm driven medication titration: Clinical pharmacists will change medications to achieve goals in hypertension, dyslipidemia and diabetes
  Monitoring: Clinical pharmacists will monitor the progress of patients in lifestyle modification and cardiac risk factor control goals
  Group support: Peer support are provided in the group setting
  Self efficacy: Patients are taught with self-monitoring skills for diabetes and blood pressure, as well as healthy cooking and practiced under supervision
Arm/Group | Pharmacist-led Group Visits | Usual Care
Number analyzed (Participants) | 117 | 133
Scores of SF-36v
  Baseline Physical Composite Summary Score | 39.2 (9.7) | 39.3 (9.8)
  13 Months Physical Composite Scores: number analyzed (Participants) | 99 | 118
  13 Months Physical Composite Scores | 39.6 (10.5) | 39.1 (9.7)
  Baseline Mental Composite Summary Score | 48.8 (11.0) | 50.4 (11.7)
  13 Months Mental Composite Summary Score: number analyzed (Participants) | 99 | 118
  13 Months Mental Composite Summary Score | 50.1 (10.5) | 51.0 (11.0)

4. Secondary Outcome: Health-care Costs to the VHA
Description: The reported values represent the "Total VHA expenditure per person". Institutional costs from health service utilization on the study patients during and 13 months after the intervention. Baseline is considered time 0.
Time Frame: 13 months (during study) and 13 months (after the study) = 26 months
Population: 117 patients randomized to Pharmacist-led Group Medical Visits. 133 patients were randomized to Usual care.
Measure: Mean (Standard Deviation); unit: United States Dollar
Arm/Group | Pharmacist-led Group Medical Visits | Usual Care
Number analyzed (Participants) | 117 | 133
United States Dollar
  baseline or time "0" | 22062 (67524) | 15200 (23812)
  Study period - 13 months prior to baseline | 4656 (31881) | 2645 (25580)
  13 months after study - study period | -1575 (30774) | 2360 (23708)
  13 months after study - 13 months before baseline: number analyzed (Participants) | 112 | 127
  13 months after study - 13 months before baseline | 4220 (31091) | 5752 (29690)

ADVERSE EVENTS:
Time Frame: 13 months of the study period
Description: Collection via monthly phone calls and face-to-face study visits
Arm/Group | Pharmacist-led Group Medical Visits | Usual Care
Serious Adverse Events (participants affected / at risk) | 38/117 | 44/133
Other Adverse Events (participants affected / at risk) | 5/117 | 7/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pharmacist-led Group Medical Visits (N=117) | Usual Care (N=133)
ER visits (General disorders) | 24 (33) | 24 (30) — Emergency room visits
hospitalization (General disorders) | 26 (40) | 21 (25) — Any cause hospitalization
Death (General disorders) | 2 (2) | 4 (4) — Any cause mortality
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pharmacist-led Group Medical Visits (N=117) | Usual Care (N=133)
Hypoglycemia, (Endocrine disorders) | 2 (117) | 1 (133) — Required unscheduled visits to the provider
Hyperglycemia (Endocrine disorders) | 3 (3) | 6 (6) — Required unscheduled visits to the provider

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No